CLINICAL TRIAL: NCT01238484
Title: Ankle Equinus Contracture Treated With Dynamic Splinting in a Randomized, Controlled Trial
Brief Title: Ankle Equinus Contracture Treated With Dynamic Splinting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Centers could not meet enrollment goals
Sponsor: Dynasplint Systems, Inc. (Industry)
Collaborators: McMurry University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010:004
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Ankle Equinus; Ankle Contracture; Diabetes Mellitus
Keywords: Ankle Equinus; Ankle contracture; Diabetes Mellitus; Dynasplint; AFD
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients in the control group will be treated with the current standard of care including shoe modification and home stretching exercises.
  Interventions: Other: Standard of care
- Experimental (Experimental): Patients assigned to the experimental group will receive the current standard of care as well as the Ankle Dorsiflexion Dynasplint.
  Interventions: Device: Dynasplint

INTERVENTIONS:
Other: Standard of care — shoe modification home stretching exercises
  Arms: Control
Device: Dynasplint — shoe modification home stretching exercises Ankle Dorsiflexion Dynasplint
  Arms: Experimental

SUMMARY:
The purpose of this study is to determine if the Ankle Dorsiflexion Dynasplint System (DS) is effective in treating contracture for patients with Ankle Equinus secondary to diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Previous Diagnosis Diabetes Mellitus
* Reduced flexibility in AROM of extension in the ankle
* Less than 10º Maximal, Active Dorsiflexion, while upright
* Impaired gait pattern

Exclusion Criteria:

* Previous surgical treatment for this pathology
* Previous surgery of the Achilles tendon or triceps surae
* Current treatment with corticosteroids
* Current treatment with Botulinium Toxin-A (Botox), lower extremity
* Current treatment Fluoroquinolones (antibiotic medication)
* Current use of muscle relaxant medications
* Fibromyalgia
* Stroke, CVA, Brain Injury, Spinal Cord Injury, or any neural pathology causing plasticity or hypertonicity
* Current participation in manual, physical therapy
* Treatment with electrical stimulation assisting ambulation (i.e. Bioness, WalkAide, Parastep, etc.)
* Preexisting open sores on foot or leg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 4 months
  The primary outcome is change in ankle range of motion

SECONDARY OUTCOMES:
Pain | 4 months
  The secondary outcome will be change in pain scale rating as reported by patient

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta Foot and Leg Clinic, Jonesboro, Georgia
  - Lopez Ankle and Foot, Fort Worth, Texas

REFERENCES:
- [Background] Van Gils CC, Roeder B. The effect of ankle equinus upon the diabetic foot. Clin Podiatr Med Surg. 2002 Jul;19(3):391-409, vi. doi: 10.1016/s0891-8422(02)00010-1. PMID 12379973
- [Background] Lavery LA, Armstrong DG, Boulton AJ; Diabetex Research Group. Ankle equinus deformity and its relationship to high plantar pressure in a large population with diabetes mellitus. J Am Podiatr Med Assoc. 2002 Oct;92(9):479-82. doi: 10.7547/87507315-92-9-479. PMID 12381796
- [Background] Armstrong DG, Boulton AJ. Continuous Internet-based activity monitoring provides a surrogate marker for nocturnal polyuria in persons with diabetes mellitus at high risk for foot ulceration. Diabet Med. 2002 Dec;19(12):1034-5. doi: 10.1046/j.1464-5491.2002.00696_2.x. No abstract available. PMID 12647847
- [Background] Dananberg HJ, Shearstone J, Guillano M. Manipulation method for the treatment of ankle equinus. J Am Podiatr Med Assoc. 2000 Sep;90(8):385-9. doi: 10.7547/87507315-90-8-385. PMID 11021048
- [Background] Lopez AA, Kalish SR, John MM, Willis FB. Reduction of Ankle Equinus Contracture Secondary to Diabetes Mellitus with Dynamic Splinting. Foot & Ankle Online Journal. 2010 3(3):13-18
- [Background] Birke JA, Patout CA Jr, Foto JG. Factors associated with ulceration and amputation in the neuropathic foot. J Orthop Sports Phys Ther. 2000 Feb;30(2):91-7. doi: 10.2519/jospt.2000.30.2.91. PMID 10693087
- [Background] Wallny T, Brackmann H, Kraft C, Nicolay C, Pennekamp P. Achilles tendon lengthening for ankle equinus deformity in hemophiliacs: 23 patients followed for 1-24 years. Acta Orthop. 2006 Feb;77(1):164-8. doi: 10.1080/17453670610045867. PMID 16534718
- [Background] Grady JF, Saxena A. Effects of stretching the gastrocnemius muscle. J Foot Surg. 1991 Sep-Oct;30(5):465-9. PMID 1783755
- [Background] Bowers AL, Castro MD. The mechanics behind the image: foot and ankle pathology associated with gastrocnemius contracture. Semin Musculoskelet Radiol. 2007 Mar;11(1):83-90. doi: 10.1055/s-2007-984418. PMID 17665354
- [Background] Mullaney MJ, McHugh MP, Tyler TF, Nicholas SJ, Lee SJ. Weakness in end-range plantar flexion after Achilles tendon repair. Am J Sports Med. 2006 Jul;34(7):1120-5. doi: 10.1177/0363546505284186. Epub 2006 Feb 13. PMID 16476917
- [Background] Chen L, Greisberg J. Achilles lengthening procedures. Foot Ankle Clin. 2009 Dec;14(4):627-37. doi: 10.1016/j.fcl.2009.08.002. PMID 19857837
- [Background] Lai J, Jones M, Willis B. Effect of Dynamic Splinting on Excessive Plantar Flexion Tone/Contracture: A Controlled, Cross-Over study. Proceedings of the 16th European Congress of Physical and Rehabilitation Medicine. Minerva Medica pubs, Italy, August 2008, pg 106-109.
- [Background] Lundequam P, Willis FB. Dynamic splinting home therapy for toe walking: a case report. Cases J. 2009 Nov 10;2:188. doi: 10.1186/1757-1626-2-188. PMID 19946498
- [Background] Sheridan L, Lopez A, Perez A, John MM, Willis FB, Shanmugam R. Plantar fasciopathy treated with dynamic splinting: a randomized controlled trial. J Am Podiatr Med Assoc. 2010 May-Jun;100(3):161-5. doi: 10.7547/1000161. PMID 20479445
- [Background] Kalish SA, Willis FB. Hallux Limitus and Dynamic Splinting: a Retrospective Series. The Foot & Ankle Online Journal 2009 Apl;2(4),1
- [Background] Huang ES, Basu A, O'Grady M, Capretta JC. Projecting the future diabetes population size and related costs for the U.S. Diabetes Care. 2009 Dec;32(12):2225-9. doi: 10.2337/dc09-0459. PMID 19940225
- [Background] Kooistra B, Dijkman B, Einhorn TA, Bhandari M. How to design a good case series. J Bone Joint Surg Am. 2009 May;91 Suppl 3:21-6. doi: 10.2106/JBJS.H.01573. PMID 19411496